CLINICAL TRIAL: NCT04095403
Title: Tarp Assisted Cooling of Hyperthermic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Riana Pryor, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003727
Record Dates: First submitted 2019-09-13; First posted 2019-09-19 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Healthy
Keywords: Heat; Cooling

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tarp assisted cooling (Experimental): Whole body cooling in a small amount of 20'C water.
  Interventions: Other: Tarp Assisted Cooling
- Passive cooling (Sham Comparator): Supine lying
  Interventions: Other: passive cooling

INTERVENTIONS:
Other: Tarp Assisted Cooling — Body cooling utilizing a tarp and water
  Arms: Tarp assisted cooling
Other: passive cooling — Supine rest.
  Arms: Passive cooling

SUMMARY:
This is a randomized controlled trial exploring the difference in cooling rates between two treatments: 1) tarp-assisted cooling and 2) the standard of care for heat stroke treatment in the wilderness.

DETAILED DESCRIPTION:
This is a randomized controlled trial exploring the difference in cooling rates between two treatments: 1) tarp-assisted cooling and 2) the standard of care for heat stroke treatment in the wilderness. 12 healthy participants (6 males, 6 females) will participate. Visit 1 will be a screening visit, consisting of informed consent followed by completion of questionnaires to determine study eligibility. Participants will have their resting vital signs (heart rate, blood pressure), height, weight, and percent body fat measured. Visits 2 and 3 will be experimental trials. Participants will complete a treadmill protocol consisting of brisk walking wearing a weighted backpack (40 lb) until core temperature reaches 40.0°C. Upon completion of exercise, participants will exit the environmental chamber and be cooled in one of two ways in a randomized, counterbalanced manner: 1) tarp-assisted cooling or 2) Standard of Care. Cooling will take place for 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Aerobic exercise at least twice weekly

Exclusion Criteria:

* History of exertional heat illness

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Cooling Rate | 20 minutes post-exercise.
  Internal body temperature reduction throughout cooling

CONTACTS AND LOCATIONS:
Overall Officials: Riana R Pryor, PhD, Principal Investigator — University at Buffalo
Locations (1):
- Center for Research and Exercise in Special Environments, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data can be shared upon request.